CLINICAL TRIAL: NCT06038188
Title: Effectiveness of a Remote 3-week Booster Intervention to Reduce Sedentary Time in Patients With Coronary Artey Disease: a Randomized Clinical Trial.
Brief Title: Remote 3-week Booster Intervention to Reduce Sedentary Time in Patients With Coronary Artey Disease
Acronym: BOOSTSITLESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NL72604.091.20; #2017T051 (Other Grant/Funding Number: senior E-Dekker grant)
Record Dates: First submitted 2023-08-30; First posted 2023-09-14 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2023-06

CONDITIONS: Coronary Artery Disease
Keywords: Cardiac rehabilitation; e-Health; Prevention; Sedentary lifestyle; Physical activity
MeSH Terms: conditions — Coronary Artery Disease; Sedentary Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The control group will receive usual care alone
- SIT LESS Booster (Experimental): The intervention group will receive usual care in combination with the remote 3-week SIT LESS Booster program.
  Interventions: Behavioral: SIT LESS Booster

INTERVENTIONS:
Behavioral: SIT LESS Booster — Patients allocated to the SIT LESS Booster group receive usual care in combination with the SIT LESS Booster program.
  The SIT LESS Booster program consists of: 1) The use of the pocket-worn activity tracker (Activ8sit). The activity tracker can be connected to an app to track the daily sitting time. Besides, the device buzzes when a person sits more than 30 consective minutes a s a reminder to stand up and move; 2) Telephone consultation (TC1) during which the researcher and patients will reactivate knowledge on the detrimental health effects of SB, discuss patients' personal goals and motivation, and collaboratively set action plans for reducing SB in the upcoming week (±20 minutes); and 3) Weekly telephone calls (TC2 and TC3) to evaluate sedentery behaviour of the preceding week (±10 minutes).
  The SIT LESS Booster will be delivered completely remote
  Arms: SIT LESS Booster

SUMMARY:
The goal of this clinical trial is to learn about the effect of a booster program aiming to lower daily sitting time (SIT LESS Booster program) compared to usual care in patient with coronary heart problems. The main question it aims to answer is: What is the effect of the SIT LESS Booster on sedentary time and physical activity levels in patient with coronary artery disease who participated in cardiac rehabilitation.

Participants will be randomized into 2 groups:

1. Control group who receives usual care;
2. SIT LESS Booster group who receives usual care + a remote 3-week SIT LESS Booster program.

Objectively measured changes in daily sitting time from pre- to post SIT LESS Booster will be compared between groups to see if participants in the SIT LESS Booster group are able to reduce daily sedentary time more compared to participants in the control group.

DETAILED DESCRIPTION:
High levels of sedentary time (ST) are observed in patients with coronary artery disease (CAD) and are associated with adverse health outcomes. Behavioural interventions targeting ST are effective in the short-term, but effects seem to diminish at long-term follow-up. Short-term (telephonic) booster programs can induce sustainable physical activity behavioural changes. However, the effects of a booster ST reduction program are unknown. Therefore, we aim to assess the effect of the SIT LESS Booster on sedentary time and physical activity levels in patient with coronary artery disease who participated in cardiac rehabilitation.

All participants took already part in a special cardiac rehabilitation program aiming to lower daily sitting time between May 2021 and April 2022. For this study, they will be randomized into 2 groups:

1. Control group who receives usual care;
2. SIT LESS Booster group who receives usual care + a remote 3-week SIT LESS Booster program.

The SIT LESS Booster program consists of:

* Telephone consultation in which the participants are informed about the negative effects of high daily sitting time, discuss personal goals to lower daily sitting time and make an action plan to reach the goals.
* Use of a pocket-worn activity tracker to get insight in their own daily sitting time. The activity tracker can be connected to a smartphone application. Besides, the activity tracker buzzes when a person sits more than 30 consecutive minutes as a reminder to stand up.
* Weekly telephone calls to discuss the progress regarding their personal sit less goals.

In both groups, daily sitting time will be measured at the start of the study and at the end of the SIT LESS Booster program using the ActivPAL.

Data analysis will be conducted using R and p-values of <0.05 will be considered statistically significant. Changes in daily ST will be compared between groups using a linear mixed model.

This trial was approved by the Medical Ethics Committee of the Radboud university medical center (NL72604.091.20)

ELIGIBILITY:
Inclusion Criteria:

• Participation in the SIT LESS intervention group of the SIT LESS study

Exclusion Criteria:

* Unable to give informed consent
* Wheelchair-bounded / not physically able to stand or walk.
* Language barrier
* Coronary arterial bypass graft surgery expected within 8 weeks after inclusion
* New York Heart Association class III or IV heart failure
* Participation in another interventional study targeting SB or PA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-08-30 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Daily Sedentary time (h/day) | Before the SIT LESS Booster program and in week 3 of the SIT LESS Booster program
  Daily sedentary time as measured with the ActivPAL during 7 days

SECONDARY OUTCOMES:
Number of prolonged sedentary bouts per day | Before the SIT LESS Booster program and in week 3 of the SIT LESS Booster program
  Daily number of prolonged sedentary bouts (>30 min/day) as measured with the ActivPAL during 7 days
Prevalence of a sitting time >9.5 h/day | Before the SIT LESS Booster program and in week 3 of the SIT LESS Booster program
  Prevalence of an average sitting time >9.5 h/day measured by the ActivPAL for 7 consective days
daily light-intensity physical activity time (h/day) | Before the SIT LESS Booster program and in week 3 of the SIT LESS Booster program
  Daily time spent in light-intensity physical activity (<3 METs) measured by the ActivPAL for 7 consective days
daily moderate-to-vigorous-intensity physical activity time (h/day) | Before the SIT LESS Booster program and in week 3 of the SIT LESS Booster program
  Daily time spent in moderate to vigorous intensity physical activity (>3 METs) measured by the ActivPAL for 7 consective days
daily step count (steps/day) | Before the SIT LESS Booster program and in week 3 of the SIT LESS Booster program
  daily step count measured by the ActivPAL for 7 consective days
Uptake of the SIT LESS Booster | from the start of recruitment (end August 2023) until 3 months later
  Number of participants participating in the SIT LESS Booster study compared to the number of eligible participants
Average wear time of the Activ8 in the SIT LESS Booster group | During the 3-week SIT LESS Booster program
  Adherence to the use of the Activ8 (wear time) measured during the intervention period in the intervention group
Number of completed telephone calls in the SIT LESS Booster group | During the 3-week SIT LESS Booster program
  Number of completed telephone calls of participants in the SIT LESS Booster group

CONTACTS AND LOCATIONS:
Overall Officials: Thijs MH Eijsvogels, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
In line with the Open Science initiative and FAIR principles, IPD will be available on reasonable request via the corresponding author.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: IPD will be availabe after publication of the results by the research team.
Access Criteria: All data will be stored in the Digital Research Environment (DRE, mydre. org), an online, cloud- based, globally available research platform. The DRE facilitates users to collaborate on research projects within the boundaries of data management regulations (General Data Protection Regulation and Good Clinical Practice compliant) in a flexible and safe way regarding security, Information and Communication Technology (ICT) infrastructure and audit trail.

REFERENCES:
- [Background] van Bakel BMA, Kroesen SH, Gunal A, Scheepmaker A, Aengevaeren WRM, Willems FF, Wondergem R, Pisters MF, Dam J, Janssen AM, de Bruin M, Hopman MTE, Thijssen DHJ, Eijsvogels TMH. Sedentary Behaviour Intervention as a Personalised Secondary Prevention Strategy (SIT LESS) for patients with coronary artery disease participating in cardiac rehabilitation: rationale and design of the SIT LESS randomised clinical trial. BMJ Open Sport Exerc Med. 2022 May 24;8(2):e001364. doi: 10.1136/bmjsem-2022-001364. eCollection 2022. PMID 35692440
- [Background] van Bakel BMA, Kroesen SH, Bakker EA, van Miltenburg RV, Gunal A, Scheepmaker A, Aengevaeren WRM, Willems FF, Wondergem R, Pisters MF, de Bruin M, Hopman MTE, Thijssen DHJ, Eijsvogels TMH. Effectiveness of an intervention to reduce sedentary behaviour as a personalised secondary prevention strategy for patients with coronary artery disease: main outcomes of the SIT LESS randomised clinical trial. Int J Behav Nutr Phys Act. 2023 Feb 14;20(1):17. doi: 10.1186/s12966-023-01419-z. PMID 36788615
- [Derived] Kroesen SH, van Bakel BMA, de Bruin M, Pisters MF, Ortega FB, Hopman MTE, Thijssen DHJ, Bakker EA, Eijsvogels TMH. A remote booster program to attenuate sedentary behaviour in patients with coronary artery disease: A Randomized Controlled Trial. Eur J Prev Cardiol. 2025 Mar 20:zwaf162. doi: 10.1093/eurjpc/zwaf162. Online ahead of print. PMID 40112182

DOCUMENTS (2):
  • Study Protocol (2023-02-28): https://cdn.clinicaltrials.gov/large-docs/88/NCT06038188/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-25): https://cdn.clinicaltrials.gov/large-docs/88/NCT06038188/SAP_001.pdf